CLINICAL TRIAL: NCT03514290
Title: Effect of Low-level Laser Therapy on Post-bleaching Sensitivity and Color Change: a Clinical, Randomized and Double-blind Study
Brief Title: Effect of Low-level Laser Therapy on Post-bleaching Sensitivity and Color Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Full professor, Universidade Federal do Para
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-003
Record Dates: First submitted 2018-03-15; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Tooth Bleaching; Low-level Laser Therapy; Dentin Sensitivity; Clinical Trial
Keywords: Laser; Color
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tooth Bleaching

STUDY DESIGN:
Intervention Model Description: Twenty-one volunteers were evaluated through the split-mouth model, so that the right and left maxillary/mandibular quadrants were randomized and allocated to one of two groups: GPLACEBO - the laser tip was positioned without the emission of light (placebo effect) + tooth bleaching with 35% hydrogen peroxide (HP); GLASER - treated with LLL + tooth bleaching with 35% HP.
Who Masked: Participant, Investigator
Masking Description: Only principal investigator performed the clinical research steps. A single evaluator performed the assessment of the dental sensitivity without knowing which treatment was applied. The volunteers evaluated in this study also did not know which hemi-arch received the LLL.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPLACEBO (Placebo Comparator): the laser tip was positioned without the emission of light (placebo effect) + tooth bleaching with 35% hydrogen peroxide (HP).
  Interventions: Other: Tooth bleaching; Other: Placebo
- GLASER (Experimental): treated with Low-lever laser + tooth bleaching with 35% hydrogen peroxide (HP).
  Interventions: Radiation: Low-lever laser; Other: Tooth bleaching

INTERVENTIONS:
Radiation: Low-lever laser — Received Low-lever laser therapy using the infrared spectrum, with a wavelength of 808 nm in its active medium AsGaAl (arsenic-gallium-aluminum), at two points: on the central of cervical and medial regions of incisors, canines and premolars in the corresponding hemi-arch. At each point, 60 J/cm2 was applied during 16 seconds with an irradiance of 3.75 W/cm² using the therapeutic visible infrared device.
  Other Names: Laserterapy
  Arms: GLASER
Other: Tooth bleaching — Three 15-minute applications of 35% hydrogen peroxide gel (Whiteness HP, FGM®, Joinville, SC, Brazil) were carried out, totaling 45 minutes in each of the four bleaching sessions, with an one-week interval between applications.
Other: Placebo — The laser tip was positioned similarly to experimental group but without light irradiation
  Arms: GPLACEBO

SUMMARY:
Objective: The objective of this clinical study was to evaluate low-level laser (LLL) therapy in tooth sensitivity and in effecting color change after in-officer bleaching treatment across three weeks of treatment.

Methods: Twenty-one volunteers were evaluated through the split-mouth model, so that the right and left maxillary/mandibular quadrants were randomized and allocated to one of two groups: GPLACEBO - the laser tip was positioned without the emission of light (placebo effect) + tooth bleaching with 35% hydrogen peroxide (HP); GLASER - treated with LLL + tooth bleaching with 35% HP. To assess tooth sensitivity, a modified visual analogue scale (VAS) was used after an evaporative stimulus (stimulated pain) and a daily pain questionnaire (unstimulated pain) was also applied. A spectrophotometer was used to measure the color. Three bleaching sessions were performed, with intervals of 7 days. Sensitivity results were tested using Friedman test for intra-group evaluation and Wilcoxon test for inter-group evaluation and ANOVA for color change.

DETAILED DESCRIPTION:
Twenty-one volunteers were evaluated through the split-mouth model, so that the right and left maxillary/mandibular quadrants were randomized and allocated to one of two groups: GPLACEBO - the laser tip was positioned without the emission of light (placebo effect) + tooth bleaching with 35% hydrogen peroxide (HP); GLASER - treated with LLL + tooth bleaching with 35% HP. To assess tooth sensitivity, a modified visual analogue scale (VAS) was used after an evaporative stimulus (stimulated pain) and a daily pain questionnaire (unstimulated pain) was also applied. A spectrophotometer was used to measure the color. Three bleaching sessions were performed, with intervals of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Do not have previous dental sensitivity
* The canine had to be shade A2 or darker.

Exclusion Criteria:

* Enamel hypoplasia
* Gingival recession
* Dentin exposure
* Visible cracks on buccal enamel
* Pulpitis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Dental sensitivity induced by office bleaching | change in baseline sensitivity at the 3rd bleaching session
  Evaporative stimulus (stimulated pain) using air jet from a triple syringe and a daily pain questionnaire (unstimulated pain). Both methods were associated with a modified visual analogue scale was used: 0 (pain absent); 1 (mild pain); 2 (moderate pain) and 3 (severe pain).

SECONDARY OUTCOMES:
Color change promoted by tooth bleaching | change in baseline color at the 3rd bleaching session
  Spectrophotometer was used to measure the color

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, Principal Investigator — Federal University of Para
Locations (1):
- Federal University of Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No